CLINICAL TRIAL: NCT00737750
Title: Phase III Study in Patients Undergoing Rehabilitation Post-Surgical Reconstruction of the Anterior Cruciate Ligament (ACL)
Brief Title: Effectiveness of Kneehab in Strengthening the Quadriceps of Patients Post Anterior Cruciate Ligament (ACL) Reconstruction
Acronym: NMES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-Medical Research, Ltd. (Industry)
Responsible Party: Prof. Hans H. Paessler, Centre for Knee and Foot Surgery, Sports Traumatology, ATOS Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BMR 04 2001A
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2008-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Neuromuscular electrical stimulation (NMES); Knee Surgery; Anterior cruciate ligament; Atrophy Prevention; Accelerated Recovery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- KH (Experimental): Kneehab is a garment integrated NMES device with multipath technology.
  Interventions: Device: Kneehab
- PS (Active Comparator): Poli-Stim, a standard NMES device, used for 3 times per day, five days per week for 12 weeks.
  Interventions: Device: Poli-Stim
- CO (Active Comparator): Control group performed voluntary muscle contractions for 20 minutes 3 times per day, 5 days per week for 12 weeks.
  Interventions: Behavioral: Control

INTERVENTIONS:
Device: Kneehab — Program of NMES 3 times per day, five days per week for 12 weeks.
  Other Names: Kneehab, neurotech
  Arms: KH
Device: Poli-Stim — Poli-Stim is standard NMES which the patients used for 20 minutes, 3 times per day, 5 days per week for 12 weeks.
  Other Names: Poli-Stim, Neurotech
  Arms: PS
Behavioral: Control — Voluntary quadriceps muscle contractions.
  Arms: CO

SUMMARY:
Prospective, controlled, randomized, single blind study in patients undergoing rehabilitation following anterior cruciate ligament reconstruction. 96 patients were randomly assigned to one of three groups. Group Group KH (Kneehab n=33)trained with a new type of garment integrated NMES for 20 minutes, 3 times per day, 5 days per week for 12 weeks; Group PS (Poli-Stim n=29) trained with standard neuromuscular electrical stimulation (NMES) for 20 minutes per day, 5 days per week for 12 weeks; Group CO (Control - n=34), which did not use muscle stimulation, performed voluntary isometric quadriceps muscle contractions. Patients receiving either form of NMES treatment were instructed to isometrically contract the quadriceps muscle voluntarily with each electrical muscle stimulation. All three groups superimposed this training schedule on the standard post-ACL reconstruction rehabilitation protocol used at the clinic.

The study design corresponded to a two-way variance analysis with three groups and 4 examination times (Baseline, 6 weeks, 12 weeks and 24 weeks post ACL reconstruction). The level of significance was set at 5%. The key indicators of the quadriceps muscle training intervention were the isokinetic strength development of the extensors of the injured leg at 90 degrees/second and 180 degrees/second and the distance achieved by participants performing the single-leg hop, the shuttle run. The target was to show a difference of 10% in the relative distance jumped for the single-leg hop and for the isokinetic strength tests and a 1.2 second difference in the time to complete the shuttle run. The target of 3 weeks was set for participants to achieve full weight-bearing capability with use of a walking aid. A comparison between the groups of the time for return to usual work activities was planned.

DETAILED DESCRIPTION:
Single center, prospective, controlled, randomized, single blind study in 96 patients following anterior crucial ligament (ACL)reconstruction to compare the effect of adding traditional NMES or garment-integrated NMES to a standard post-surgery rehabilitation program. In both cases the NMES was superimposed on isometric voluntary muscle contractions.

ELIGIBILITY:
Inclusion Criteria:

* Persons who had surgical reconstruction of the anterior cruciate ligament
* Persons with additional treatment of minor miniscal defects
* Persons who were willing and able to provide Informed Consent

Exclusion Criteria:

* Persons who had multi-ligament reconstruction
* ACL patients with a microfracture or extra burden on the knee
* Persons who registered pain above level 3 on the IKDC subjective evaluation pain scale questions, 3 days after surgery
* Participants in a volunteer study within the previous ninety (90) days
* Persons with serious cardiac arrhythmias or other implanted devices
* Persons with cardiac pacemakers
* Persons with neurological or psychiatric disorders
* Persons who are pregnant or breastfeeding
* Intake of drugs that interfere with the neuromuscular system
* Persons with epilepsy
* Any condition or history which in the opinion of the Principal Investigator might increase the risk to an individual or interfere with the evaluation of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2005-04; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Isokinetic strength test of extension of the injured leg. Relative strength extension ratio (injured/uninjured). Distance of the jump achieved in the single leg hop and the time to achieve the shuttle run. | 12 weeks Intervention + Outcomes at 24 Weeks

SECONDARY OUTCOMES:
Strength test of flexors of the knee joint and 5 tests of coordination of proprioceptions (triple hop; side-step; carioca; timed hop and cross-over hop). | 12 weeks Intervention + Outcomes at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans H Paessler, FRCSed, Principal Investigator — Centre for Knee and Foot Surgery Sports Traumatology, ATOS Clinic, Heidelberg, Germany
Locations (1):
- ATOS Clinic, Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Andersson C, Odensten M, Gillquist J. Knee function after surgical or nonsurgical treatment of acute rupture of the anterior cruciate ligament: a randomized study with a long-term follow-up period. Clin Orthop Relat Res. 1991 Mar;(264):255-63. PMID 1997243
- [Background] Barber SD, Noyes FR, Mangine RE, McCloskey JW, Hartman W. Quantitative assessment of functional limitations in normal and anterior cruciate ligament-deficient knees. Clin Orthop Relat Res. 1990 Jun;(255):204-14. PMID 2347154
- [Background] Bax L, Staes F, Verhagen A. Does neuromuscular electrical stimulation strengthen the quadriceps femoris? A systematic review of randomised controlled trials. Sports Med. 2005;35(3):191-212. doi: 10.2165/00007256-200535030-00002. PMID 15730336
- [Background] Barrack RL, Skinner HB, Buckley SL. Proprioception in the anterior cruciate deficient knee. Am J Sports Med. 1989 Jan-Feb;17(1):1-6. doi: 10.1177/036354658901700101. PMID 2929825
- [Background] Barrett DS. Proprioception and function after anterior cruciate reconstruction. J Bone Joint Surg Br. 1991 Sep;73(5):833-7. doi: 10.1302/0301-620X.73B5.1894677.
- [Background] Beynnon BD, Fleming BC, Johnson RJ, Nichols CE, Renstrom PA, Pope MH. Anterior cruciate ligament strain behavior during rehabilitation exercises in vivo. Am J Sports Med. 1995 Jan-Feb;23(1):24-34. doi: 10.1177/036354659502300105. PMID 7726347
- [Background] Currier DP, Ray JM, Nyland J, Rooney JG, Noteboom JT, Kellogg R. Effects of electrical and electromagnetic stimulation after anterior cruciate ligament reconstruction. J Orthop Sports Phys Ther. 1993 Apr;17(4):177-84. doi: 10.2519/jospt.1993.17.4.177. PMID 8467342
- [Background] Delitto A, Rose SJ, McKowen JM, Lehman RC, Thomas JA, Shively RA. Electrical stimulation versus voluntary exercise in strengthening thigh musculature after anterior cruciate ligament surgery. Phys Ther. 1988 May;68(5):660-3. doi: 10.1093/ptj/68.5.660. PMID 3258994
- [Background] Draganich LF, Vahey JW. An in vitro study of anterior cruciate ligament strain induced by quadriceps and hamstrings forces. J Orthop Res. 1990 Jan;8(1):57-63. doi: 10.1002/jor.1100080107. PMID 2293634
- [Background] Draper V, Ballard L. Electrical stimulation versus electromyographic biofeedback in the recovery of quadriceps femoris muscle function following anterior cruciate ligament surgery. Phys Ther. 1991 Jun;71(6):455-61; discussion 461-4. doi: 10.1093/ptj/71.6.455. PMID 2034708
- [Background] Eastlack ME, Axe MJ, Snyder-Mackler L. Laxity, instability, and functional outcome after ACL injury: copers versus noncopers. Med Sci Sports Exerc. 1999 Feb;31(2):210-5. doi: 10.1097/00005768-199902000-00002. PMID 10063808
- [Background] Engstrom B, Gornitzka J, Johansson C, Wredmark T. Knee function after anterior cruciate ligament ruptures treated conservatively. Int Orthop. 1993;17(4):208-13. doi: 10.1007/BF00194180. PMID 8407034
- [Background] Fitzgerald GK, Lephart SM, Hwang JH, Wainner RS. Hop tests as predictors of dynamic knee stability. J Orthop Sports Phys Ther. 2001 Oct;31(10):588-97. doi: 10.2519/jospt.2001.31.10.588. PMID 11665746
- [Background] Fitzgerald GK, Piva SR, Irrgang JJ. A modified neuromuscular electrical stimulation protocol for quadriceps strength training following anterior cruciate ligament reconstruction. J Orthop Sports Phys Ther. 2003 Sep;33(9):492-501. doi: 10.2519/jospt.2003.33.9.492. PMID 14524508
- [Background] Havlik E, Haber P, Klein G, Roggla G, Bergmann H. Increased 137caesium whole body radioactivity in high-performance athletes. Int J Sports Med. 1990 Feb;11(1):37-40. doi: 10.1055/s-2007-1024759. PMID 2108095
- [Background] Gobbi A, Tuy B, Mahajan S, Panuncialman I. Quadrupled bone-semitendinosus anterior cruciate ligament reconstruction: a clinical investigation in a group of athletes. Arthroscopy. 2003 Sep;19(7):691-9. doi: 10.1016/s0749-8063(03)00685-6. PMID 12966375
- [Background] Hefti F, Muller W, Jakob RP, Staubli HU. Evaluation of knee ligament injuries with the IKDC form. Knee Surg Sports Traumatol Arthrosc. 1993;1(3-4):226-34. doi: 10.1007/BF01560215. PMID 8536037
- [Background] Hehl G, Hoellen I, Wissmeyer T, Ziegler U. [Isokinetic muscle training with high motion speeds in the rehabilitation following surgical treatment of fresh anterior cruciate rupture]. Z Orthop Ihre Grenzgeb. 1995 Jul-Aug;133(4):306-10. doi: 10.1055/s-2008-1039797. German. PMID 7571796
- [Background] Jarvela T, Kannus P, Latvala K, Jarvinen M. Simple measurements in assessing muscle performance after an ACL reconstruction. Int J Sports Med. 2002 Apr;23(3):196-201. doi: 10.1055/s-2002-23171. PMID 11914983
- [Background] Keays SL, Bullock-Saxton J, Keays AC, Newcombe P. Muscle strength and function before and after anterior cruciate ligament reconstruction using semitendonosus and gracilis. Knee. 2001 Oct;8(3):229-34. doi: 10.1016/s0968-0160(01)00099-0. PMID 11706731
- [Background] Keays SL, Bullock-Saxton JE, Newcombe P, Keays AC. The relationship between knee strength and functional stability before and after anterior cruciate ligament reconstruction. J Orthop Res. 2003 Mar;21(2):231-7. doi: 10.1016/S0736-0266(02)00160-2. PMID 12568953
- [Background] Kramer J, Nusca D, Fowler P, Webster-Bogaert S. Knee flexor and extensor strength during concentric and eccentric muscle actions after anterior cruciate ligament reconstruction using the semitendinosus tendon and ligament augmentation device. Am J Sports Med. 1993 Mar-Apr;21(2):285-91. doi: 10.1177/036354659302100220. PMID 8465926
- [Background] Kvist J, Karlberg C, Gerdle B, Gillquist J. Anterior tibial translation during different isokinetic quadriceps torque in anterior cruciate ligament deficient and nonimpaired individuals. J Orthop Sports Phys Ther. 2001 Jan;31(1):4-15. doi: 10.2519/jospt.2001.31.1.4. PMID 11204794
- [Background] Lieber RL, Silva PD, Daniel DM. Equal effectiveness of electrical and volitional strength training for quadriceps femoris muscles after anterior cruciate ligament surgery. J Orthop Res. 1996 Jan;14(1):131-8. doi: 10.1002/jor.1100140121. PMID 8618155
- [Background] Chow GK, Streem SB. Extracorporeal lithotripsy. Update on technology. Urol Clin North Am. 2000 May;27(2):315-22. doi: 10.1016/s0094-0143(05)70260-3. PMID 10778473
- [Background] Morrissey MC, Brewster CE, Shields CL Jr, Brown M. The effects of electrical stimulation on the quadriceps during postoperative knee immobilization. Am J Sports Med. 1985 Jan-Feb;13(1):40-5. doi: 10.1177/036354658501300107. PMID 3872083
- [Background] Noyes FR, Mooar PA, Matthews DS, Butler DL. The symptomatic anterior cruciate-deficient knee. Part I: the long-term functional disability in athletically active individuals. J Bone Joint Surg Am. 1983 Feb;65(2):154-62. doi: 10.2106/00004623-198365020-00003. No abstract available. PMID 6687391
- [Background] Noyes FR, Matthews DS, Mooar PA, Grood ES. The symptomatic anterior cruciate-deficient knee. Part II: the results of rehabilitation, activity modification, and counseling on functional disability. J Bone Joint Surg Am. 1983 Feb;65(2):163-74. doi: 10.2106/00004623-198365020-00004. No abstract available. PMID 6822580
- [Background] Nyland J, Caborn DN, Rothbauer J, Kocabey Y, Couch J. Two-year outcomes following ACL reconstruction with allograft tibialis anterior tendons: a retrospective study. Knee Surg Sports Traumatol Arthrosc. 2003 Jul;11(4):212-8. doi: 10.1007/s00167-003-0371-x. Epub 2003 Jun 19. PMID 12827225
- [Background] Oshimo TA, Greene TA, Jensen GM, Lopopolo RB. The effect of varied hip angles on the generation of internal tibial rotary torque. Med Sci Sports Exerc. 1983;15(6):529-34. PMID 6656564
- [Background] Parker MG, Bennett MJ, Hieb MA, Hollar AC, Roe AA. Strength response in human femoris muscle during 2 neuromuscular electrical stimulation programs. J Orthop Sports Phys Ther. 2003 Dec;33(12):719-26. doi: 10.2519/jospt.2003.33.12.719. PMID 14743985
- [Background] Paessler HH, Mastrokalos DS. Anterior cruciate ligament reconstruction using semitendinosus and gracilis tendons, bone patellar tendon, or quadriceps tendon-graft with press-fit fixation without hardware. A new and innovative procedure. Orthop Clin North Am. 2003 Jan;34(1):49-64. doi: 10.1016/s0030-5898(02)00070-6. PMID 12735201
- [Background] Paillard T. Combined application of neuromuscular electrical stimulation and voluntary muscular contractions. Sports Med. 2008;38(2):161-77. doi: 10.2165/00007256-200838020-00005. PMID 18201117
- [Background] Paillard T, Noe F, Passelergue P, Dupui P. Electrical stimulation superimposed onto voluntary muscular contraction. Sports Med. 2005;35(11):951-66. doi: 10.2165/00007256-200535110-00003. PMID 16271009
- [Background] Petschnig R, Baron R, Albrecht M. The relationship between isokinetic quadriceps strength test and hop tests for distance and one-legged vertical jump test following anterior cruciate ligament reconstruction. J Orthop Sports Phys Ther. 1998 Jul;28(1):23-31. doi: 10.2519/jospt.1998.28.1.23. PMID 9653687
- [Background] Renstrom P, Arms SW, Stanwyck TS, Johnson RJ, Pope MH. Strain within the anterior cruciate ligament during hamstring and quadriceps activity. Am J Sports Med. 1986 Jan-Feb;14(1):83-7. doi: 10.1177/036354658601400114. PMID 3752352
- [Background] Rudolph KS, Axe MJ, Snyder-Mackler L. Dynamic stability after ACL injury: who can hop? Knee Surg Sports Traumatol Arthrosc. 2000;8(5):262-9. doi: 10.1007/s001670000130. PMID 11061293
- [Background] Segawa H, Omori G, Koga Y, Kameo T, Iida S, Tanaka M. Rotational muscle strength of the limb after anterior cruciate ligament reconstruction using semitendinosus and gracilis tendon. Arthroscopy. 2002 Feb;18(2):177-82. doi: 10.1053/jars.2002.29894. PMID 11830812
- [Background] Sekiya I, Muneta T, Ogiuchi T, Yagishita K, Yamamoto H. Significance of the single-legged hop test to the anterior cruciate ligament-reconstructed knee in relation to muscle strength and anterior laxity. Am J Sports Med. 1998 May-Jun;26(3):384-8. doi: 10.1177/03635465980260030701. PMID 9617400
- [Background] Shelburne KB, Pandy MG. A musculoskeletal model of the knee for evaluating ligament forces during isometric contractions. J Biomech. 1997 Feb;30(2):163-76. doi: 10.1016/s0021-9290(96)00119-4. PMID 9001937
- [Background] Snyder-Mackler L, Ladin Z, Schepsis AA, Young JC. Electrical stimulation of the thigh muscles after reconstruction of the anterior cruciate ligament. Effects of electrically elicited contraction of the quadriceps femoris and hamstring muscles on gait and on strength of the thigh muscles. J Bone Joint Surg Am. 1991 Aug;73(7):1025-36. PMID 1874764
- [Background] Snyder-Mackler L, Delitto A, Bailey SL, Stralka SW. Strength of the quadriceps femoris muscle and functional recovery after reconstruction of the anterior cruciate ligament. A prospective, randomized clinical trial of electrical stimulation. J Bone Joint Surg Am. 1995 Aug;77(8):1166-73. doi: 10.2106/00004623-199508000-00004. PMID 7642660
- [Background] Stevens JE, Mizner RL, Snyder-Mackler L. Neuromuscular electrical stimulation for quadriceps muscle strengthening after bilateral total knee arthroplasty: a case series. J Orthop Sports Phys Ther. 2004 Jan;34(1):21-9. doi: 10.2519/jospt.2004.34.1.21. PMID 14964588
- [Background] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Background] Vanderthommen M, Crielaard JM. [Muscle electric stimulation in sports medicine]. Rev Med Liege. 2001 May;56(5):391-5. French. PMID 11475938
- [Background] Viola RW, Sterett WI, Newfield D, Steadman JR, Torry MR. Internal and external tibial rotation strength after anterior cruciate ligament reconstruction using ipsilateral semitendinosus and gracilis tendon autografts. Am J Sports Med. 2000 Jul-Aug;28(4):552-5. doi: 10.1177/03635465000280041801. PMID 10921649
- [Background] Wilk KE, Romaniello WT, Soscia SM, Arrigo CA, Andrews JR. The relationship between subjective knee scores, isokinetic testing, and functional testing in the ACL-reconstructed knee. J Orthop Sports Phys Ther. 1994 Aug;20(2):60-73. doi: 10.2519/jospt.1994.20.2.60. PMID 7920603